CLINICAL TRIAL: NCT06185049
Title: Transdiagnostic Selective Preventive Intervention for At-risk Adolescents With Booster Sessions.
Brief Title: Selective Prevention Transdiagnostic Intervention for At-risk Adolescents With Booster Sessions. (PROCARE+ 2.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other); University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, LuisJoaquin Garcia-Lopez, Professor, University of Jaén
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: UJA_PROARE+ 2.0
Record Dates: First submitted 2023-12-07; First posted 2023-12-29 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Anxiety Disorders and Symptoms Depressive Symptoms; Risk Factors (Rejection, Bullying/Cyberbullying, Addictions, Healthy Lifestyle Habits, Exam Stress Management, Ecoanxiety, Expressed Emotion)
Keywords: ADOLESCENCE; TRANSDIAGNOSTIC SELECTIVE PREVENTION; RISK FACTOR; REJECTION, BULLYING/CYBERBULLYING; ADDICTIONS; HEALTHY LIFESTYLE HABITS; ECOANXIETY; EXAM STRESS; EXPRESSED EMOTION
MeSH Terms: conditions — Anxiety Disorders; Depression; Rejection, Psychology; Bullying; Cyberbullying; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: The effects of an intervention with two booster sessions will be evaluated in parallel with an intervention that only has one booster session and with an intervention without booster sessions.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PROCARE+ (Core intervention with add-on modules) and two booster sessions, at 6 and 12 months (Experimental): In addition to core UP-A preventive intervention, PROCARE + will apply an innovative personalized medicine approach by adding specific modules according to the risk factor evidenced by adolescents. Different modules will be suited for the stratified groups in a more personalized format. Add-on young-focused modules would include: rejection, bullying/cyberbullying, addictions, healthy lifestyle habits, exam stress management, ecoanxiety, parental expressed emotion. Two booster sessions would be included (at 6 and 12 months).
  Interventions: Behavioral: PROCARE+ (Core intervention with add-on modules) and two booster sessions.
- PROCARE+ (Core intervention with add-on modules) and a booster session at 6 months. (Experimental): In addition to core UP-A preventive intervention, PROCARE + will apply an innovative personalized medicine approach by adding specific modules according to the risk factor evidenced by adolescents. Different modules will be suited for the stratified groups in a more personalized format. Add-on young-focused modules would include: rejection, bullying/cyberbullying, addictions, healthy lifestyle habits, exam stress management, ecoanxiety, parental expressed emotion. A booster sessions would be included at 6 months.
  Interventions: Behavioral: PROCARE+ (Core intervention with add-on modules) and one booster session
- PROCARE+ (Core intervention with add-on modules) without booster sessions (Experimental): In addition to core UP-A preventive intervention, PROCARE + will apply an innovative personalized medicine approach by adding specific modules according to the risk factor evidenced by adolescents. Different modules will be suited for the stratified groups in a more personalized format. Add-on young-focused modules would include: rejection, bullying/cyberbullying, addictions, healthy lifestyle habits, exam stress management, ecoanxiety, parental expressed emotion. Only follow-up would be conducted up to 12 months.
  Interventions: Behavioral: PROCARE+ (Core intervention with add-on modules) without booster sessions.

INTERVENTIONS:
Behavioral: PROCARE+ (Core intervention with add-on modules) and two booster sessions. — The modules will primarily involve therapeutic sessions aimed at equipping adolescents with strategies for addressing risky situations, including enhancing their communication skills and developing coping mechanisms for stress management. The group sessions will also incorporate education on the importance of open discussions about thoughts, emotions, and behavior as integral components of emotional well-being, with a strong focus on offering support tailored to the identified risk factors. It will include two booster sessions at 6 and 12 months into the intervention.
  Other Names: PROCARE+ two booster sessions.
  Arms: PROCARE+ (Core intervention with add-on modules) and two booster sessions, at 6 and 12 months
Behavioral: PROCARE+ (Core intervention with add-on modules) and one booster session — The modules will primarily involve therapeutic sessions aimed at equipping adolescents with strategies for addressing risky situations, including enhancing their communication skills and developing coping mechanisms for stress management. The group sessions will also incorporate education on the importance of open discussions about thoughts, emotions, and behavior as integral components of emotional well-being, with a strong focus on offering support tailored to the identified risk factors. It will include abooster sessions at 6 months into the intervention.
  Other Names: PROCARE+ one booster session
  Arms: PROCARE+ (Core intervention with add-on modules) and a booster session at 6 months.
Behavioral: PROCARE+ (Core intervention with add-on modules) without booster sessions. — The modules will primarily involve therapeutic sessions aimed at equipping adolescents with strategies for addressing risky situations, including enhancing their communication skills and developing coping mechanisms for stress management. The group sessions will also incorporate education on the importance of open discussions about thoughts, emotions, and behavior as integral components of emotional well-being, with a strong focus on offering support tailored to the identified risk factors.
  Other Names: PROCARE+ without booster sessions
  Arms: PROCARE+ (Core intervention with add-on modules) without booster sessions

SUMMARY:
Emotional disorders such as anxiety and depression are significantly underdiagnosed and undertreated, even though they are some of the most prevalent mental health conditions, especially among young individuals. Approximately 50% of mental health disorders manifest by the age of 14, and around 75% appear by the age of 24, underscoring the critical importance of addressing these issues during adolescence. Unfortunately, during this developmental stage, early warning signs and even fully developed clinical conditions often go unnoticed, undiagnosed, and untreated.

Nonetheless, there is a lack of established, evidence-backed procedures aimed at reaching out to adolescents at risk of developing emotional disorders. Urgently required is a fundamental shift in our approach by creating intervention protocols that allow for the early identification and treatment of at-risk adolescents, thus averting the potential development of severe mental health disorders as they mature. The selective prevention of mental health issues is a crucial element in assisting at-risk adolescents in flourishing before emotional disorders progress. To address this gap, PROCARE+ was conceived as a modularized selective prevention program for adolescents aged 12 to 18 years. Using a personalized medicine approach, PROCARE+ successfully allowed for the adaptation of intervention protocols according to the specific needs of each individual, while also identifying vulnerable individuals based on risk factors. This research aims to maximize and extend the impact on the adolescent population in the post-COVID-19 pandemic stage and will analyze the effectiveness of implementing booster sessions. PROCARE + stratifies adolescents based on their risk and resilience status and will deliver, alongside a core intervention, new specific add-on modules designed to address risk factors identified by adolescents: : 1) Situations of rejection, bullying, and cyberbullying; 2) Addiction to new technologies such as video games or mobile phones and other substances like alcohol, tobacco, and drugs; 3) Improvement of healthy lifestyle habits related to nutrition, sleep, and physical activity; 4) Enhancement of stress-related situations: Ecoanxiety or exam-related anxiety; and 5) Improvement of parent-child relationships and situations of high expressed emotion (parent module).

In addition, the study of booster sessions will be further explored to maintain the results following the initial intervention (which is based on core and additional modules according to identified risk factors). To achieve this, a randomized controlled trial with three conditions will be conducted. Adolescents will be assigned to different experimental groups with or without booster sessions in order to increase the effectiveness of the intervention. The objective is to reduce the impact of risk factors and enhance protective factors, ultimately leading to lasting positive outcomes for adolescents. It will combine quantitative analyses, with a special focus on vulnerable groups in a disaggregated approach by sex, gender, sexual orientation, and socioeconomic status. The PROCARE project is expected to have a significant impact. Its outcomes will continue to contribute to the identification and preventive treatment of adolescents at risk of emotional mental disorders at an early stage, before they incur personal, social, and economic costs. This aims to provide new data to help improve personalized preventive medicine. It will be designed to be an acceptable, scalable, and sustainable selective prevention program, striving to increase its effectiveness beyond the context of the COVID-19 pandemic, ultimately contributing to the prevention and reduction of the prevalence of mental disorders in young people.

DETAILED DESCRIPTION:
The general objective of this research is to maximize the benefits of PRCARE+ and assess the effectiveness of implementing booster sessions following the personalized, preventive-selective transdiagnostic intervention in adolescents aged 12 to 18 years.

The core intervention is based on the Unified Protocol for the transdiagnostic treatment of emotional disorders in adolescents (UP-A), which has already demonstrated its effectiveness in the United States but, in this case, adapted for selective prevention purposes. New, enhanced specific modules are provided to address the risk factors identified by the adolescents themselves. Based on the prior stratification of adolescents according to risk and resilience factors, additional specific modules are offered to strengthen emotional regulation, resilience, and coping capacity. Special attention is paid to the effects of booster sessions that allow for the maintenance of intervention outcomes over time. All of this is accomplished through a sequenced approach to skill development, resilience, and explicit implementation guidelines. It is culturally adapted to be acceptable, scalable, and sustainable, contributing to the promotion of emotional mental health in young people.

The specific objectives of this research are as follows:

To identify adolescents at risk of emotional difficulties through a comprehensive analysis of risk and resilience factors. The personalized medicine approach will enable the team to tailor additional intervention modules according to the specific needs of each individual, as well as to determine which risk factors are the best indicators for identifying at-risk youth and/or indicators of program effectiveness.

To enhance the transdiagnostic, preventive-selective, and personalized PROCARE+ intervention for adolescents at risk of developing mental health problems such as anxiety and depression. The preventive program will be adapted from the UP-A protocol for the clinical population, and new additional modules will be applied based on the presented risk factors. This will be implemented through a personalized telemedicine approach. The project has the support of a strong External Advisory Board (EAB): Asociación Española de Ayuda Mutua contra Fobia Social y Trastornos de Ansiedad (AMTAES), Federación Estatal de Lesbianas, Gais, Trans y Bisexuales (FELGTB), Instituto de la Juventud (INJUVE/Ministerio de Asuntos Sociales y Agenda 2030 de España) y Confederación de Organizaciones de Psicopedagogía y Orientación de España (COPOE), Consejo de la juventud de España (CJE).

To demonstrate the cost-effectiveness of booster sessions by designing a trial with three conditions: 1) PROCARE + (Core intervention with add-on modules) and two booster sessions, at 6 and 12 months; 2) PROCARE + (Core intervention with add-on modules) and one booster session, at 6 months; 3) PROCARE + (Core intervention with add-on modules) without booster sessions. All conditions will include baseline, post-test, 6-month, and one-year follow-ups. PROCARE will adhere to internationally adopted guidelines to maximize the reliability of results in preventive trials. The evaluation will combine quantitative and qualitative methods, and the analysis of findings will be conducted: (a) qualitatively, (b) quantitatively, and (c) disaggregated by gender, examining differences between boys and girls and data intersecting with gender (cultural gender norms and emotion regulation skills) that can help explain these differences.

METHODOLOGY The methodology was designed in response to current trends in selective prevention and personalized medicine. The work plan for this research will be divided into three interconnected stages.: Assessment and Stratification; Intervention; and Booster and Follow-up. First, to identify adolescents at risk of experiencing emotional disorders (anxiety and depression), the following questionnaires will be administered to the adolescents: Strengths and Difficulties Questionnaire (SDQ) to assess adolescents at risk of emotional disorders, the Connor-Davidson Resilience Scale (CD-RISC) to assess resilience, the Revised Child Anxiety and Depression Scale-30 (RCADS-30) to detect the presence/absence of emotional symptomatology, the Kidscreen-10 scale for self-reported quality of life assessment, the Difficulties in Emotion Regulation Scale (DERS) as a measure of emotional regulation, and the Willingness and Action Measure for Children and Adolescents (WAM-C/A) as a measure of psychological flexibility. Additionally, potential risk factors will be collected from adolescents and parents through the Climate Anxiety Scale (CAS) by Clayton and Karazsia; Exam Anxiety Questionnaire adapted for Secondary Education (CAEX-A); Cyberbullying and bullying scale; Structured Interview for the Assessment of Expressed Emotion: Child version (E5cv); Video Game Addiction Scale for Adolescents (GASA); Short Version Smartphone Addiction Scale (SAS-SV). These factors will be used for stratification and the adaptation of additional intervention modules according to the specific needs of each subject: (i)to identify individuals at risk and define short- and long-term mechanisms of action for the transdiagnostic, preventive-selective, and personalized PROCARE+ intervention. The researchers will test the effects of booster sessions on the maintenance of the outcomes of a selective preventive intervention using a randomized clinical trial and a personalized medicine approach, with a focus on risk factors and vulnerable youth (refugees, immigrants, or national, ethnic, linguistic, religious, and sexual minorities).

IMPACT The need to prioritize mental health on the public health agenda has been increasingly recognized over the past decades. he results of the research will have a significant impact, ultimately contributing to increasing understanding of the underlying mechanisms of selective prevention of mental disorders in young people and the maintenance of these effects. These problems are extensive, enduring, and of great magnitude, imposing a range of costs on individuals, families, and communities. Prevention will lead to the reduction of personal, social, and economic costs.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from adolescent and legal guardian
* able to attend prevention modules on his/her own
* Strengths and Difficulties Questionnaire "unlikely" or "possible diagnoses"
* score on Connor-Davidson Resilience Scale as low or medium resilient,
* score below cut-off for Revised Child Anxiety and Depression Scale-30
* evidence of risk factors (social exclusion, stress-related situations, unhealthy lifestyle habits, parental-child interaction)
* absence of anxiety and/or mood disorders
* not receiving psychological or psychiatric treatment
* not presenting acute suicidality and (9) absence of neurodevelopmental disorders.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The Strengths and Difficulties Questionnaire SDQ | Baseline to 12 months after start of interventions]
  The study's primary outcome was self-reported risk and protective factors level of emotional disorders as assessed by Strengths and Difficulties Questionnaire (SDQ).
  Only 5 items of the emotional problems subscale of the self-reported version for adolescents (Self-Reported SDQ) was used. And 5 items of the emotional problems subscale of the parent version (Parent SDQ). Items with Likert-type response format scored from 0 to 2. Higher scores mean a worse outcome.
Resilience | Baseline to 12 months after start of interventions]
  Self-reported resilience, as measured by Connor-Davidson Resilience Scale (CD-RISC-10).10 items with a Likert-type response format from 0 to 4. Total scores range from 0 to 40. Higher scores mean a better outcome.
Health-related quality of life | Baseline to 12 months after start of interventions]
  Self-reported changes in health-related quality of life as assessed by self-reported changes in health-related quality of life as assessed by KIDSCREEN-10. This instrument contains 10 items with a Likert-type response form ranging from 1 to 4. Total scores range from 10 to 40. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Emotion regulation skills | Baseline to 12 months after start of interventions]
  Emotion regulation skills as assessed by Difficulties in Emotion Regulation Scale (DERS-36), It has 36 items with a Likert-type response format ranging from 0 to 4. Total scores range from 36 to 144. Higher scores mean a worse outcome.
Psychological flexibility | Baseline to 12 months after start of interventions]
  Psychological flexibility as assessed by Willingness and Action Measure for Children and Adolescents (WAM-C/A). It has 14 items with Likert-type response format scored from 0 to 4. Total scores range from 0 to 56. Higher scores mean a better outcome.
Self-reported anxiety and mood symptomatology | Baseline to 12 months after start of interventions]
  The study's primary outcome was self-reported anxiety and mood symptomatology as assessed by Revised Child Anxiety Depression Scale (RCADS-30). It is a brief version consisting of 30 items with Likert-type responses scored from 0 to 3. Total scores range from 0 to 90. Higher scores mean a worse outcome.

OTHER OUTCOMES:
Ecoanxiety | Baseline to 12 months after start of interventions]
  Climate Anxiety Scale (CAS) by Clayton and Karazsia (2020). Assesses climate anxiety as a psychological response to climate change. It has 22 Likert-type items with 5 response options (1 to 5).
Exam anxiety | Baseline to 12 months after start of interventions]
  Exam Anxiety Questionnaire adapted for Secondary Education (CAEX-A). The 6 items with the highest factorial load from the original scale are used (2 from the cognitive subscale, 2 from the physiological subscale, and 2 from the behavioral subscale). The response format is Likert scale from 0 to 4.
Social exclusion | Baseline to 12 months after start of interventions]
  Cyberbullying and bullying scale. It has 19 items. The response format is Likert-type from 0 to 4 (''never'', ''sometimes'', ''quite often'' and ''always"), indicating the frequency in which the participant has been (cyber) victimized during the last year.
Parental-child interaction | Baseline to 12 months after start of interventions]
  Structured Interview for the Assessment of Expressed Emotion: Child version (E5cv) Five-item structured interview with five response options, ranging from 1 to 5.
video game addiction | Baseline to 12 months after start of interventions]
  Video Game Addiction Scale for Adolescents (GASA): This questionnaire allows for the assessment of problematic console use and video game addiction. It consists of 7 items on a Likert scale (1 to 5).
problematic mobile phone use | Baseline to 12 months after start of interventions]
  Short Version Smartphone Addiction Scale (SAS-SV): This scale assesses problematic mobile phone use, which leads to dependency patterns and, in addition, negative consequences. It consists of 10 items on a Likert scale (1 to 6)."
Health and lifestyle habits | Baseline to 12 months after start of interventions]
  A short 9-question questionnaire was created ad-hoc to detect different problems related to health and lifestyle habits

CONTACTS AND LOCATIONS:
Overall Officials: LuisJoaquin Garcia-Lopez, PhD, Principal Investigator — University of Jaen
Locations (1):
- University of Jaen, Jaén, Jaen, Spain

REFERENCES:
- [Background] Garcia-Escalera J, Valiente RM, Sandin B, Ehrenreich-May J, Prieto A, Chorot P. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) Adapted as a School-Based Anxiety and Depression Prevention Program: An Initial Cluster Randomized Wait-List-Controlled Trial. Behav Ther. 2020 May;51(3):461-473. doi: 10.1016/j.beth.2019.08.003. Epub 2019 Aug 14. PMID 32402261
- [Background] Sandin B, Garcia-Escalera J, Valiente RM, Espinosa V, Chorot P. Clinical Utility of an Internet-Delivered Version of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (iUP-A): A Pilot Open Trial. Int J Environ Res Public Health. 2020 Nov 10;17(22):8306. doi: 10.3390/ijerph17228306. PMID 33182711
- [Background] Levin L, Henderson HA, Ehrenreich-May J. Interpersonal predictors of early therapeutic alliance in a transdiagnostic cognitive-behavioral treatment for adolescents with anxiety and depression. Psychotherapy (Chic). 2012 Jun;49(2):218-230. doi: 10.1037/a0028265. PMID 22642525
- [Background] Queen AH, Barlow DH, Ehrenreich-May J. The trajectories of adolescent anxiety and depressive symptoms over the course of a transdiagnostic treatment. J Anxiety Disord. 2014 Aug;28(6):511-21. doi: 10.1016/j.janxdis.2014.05.007. Epub 2014 Jun 2. PMID 24960439
- [Background] Bilek EL, Ehrenreich-May J. An open trial investigation of a transdiagnostic group treatment for children with anxiety and depressive symptoms. Behav Ther. 2012 Dec;43(4):887-97. doi: 10.1016/j.beth.2012.04.007. Epub 2012 May 1. PMID 23046789
- [Background] Ehrenreich-May J, Rosenfield D, Queen AH, Kennedy SM, Remmes CS, Barlow DH. An initial waitlist-controlled trial of the unified protocol for the treatment of emotional disorders in adolescents. J Anxiety Disord. 2017 Mar;46:46-55. doi: 10.1016/j.janxdis.2016.10.006. Epub 2016 Oct 17. PMID 27771133
- [Background] Vivas-Fernandez M, Garcia-Lopez LJ, Piqueras JA, Muela-Martinez JA, Canals-Sans J, Espinosa-Fernandez L, Jimenez-Vazquez D, Diaz-Castela MDM, Morales-Hidalgo P, Rivera M, Ehrenreich-May J. Randomized controlled trial for selective preventive transdiagnostic intervention for adolescents at risk for emotional disorders. Child Adolesc Psychiatry Ment Health. 2023 Jun 23;17(1):77. doi: 10.1186/s13034-023-00616-9. PMID 37353831